CLINICAL TRIAL: NCT04508608
Title: Scintigraphic Evaluation of Contractile and Coronary Reserve in Patients With Ischemic Cardiomyopathy
Acronym: SciCoRIC
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: SciCoRIC; АААА-А15-115123110026-3 (Other: Cardiology Research Institute, Tomsk NRMC)
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2020-10

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Ischemic Cardiomyopathy; Single photon emission computed tomography; Gated blood pool SPECT; Coronary flow reserve; Prognosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ischemic cardiomyopathy group - 1 (ICM-1): Inclusion criteria:
  1. History of myocardial infarction (MI) or revascularization (CABG or PCI);
  2. > 75% stenosis of left main or proximal left anterior descending artery (LAD) and/ or stenosis of > 75% of ≥2 epicardial vessels (based on coronary angiography (CA) data);
  3. LV ejection fraction (EF) <40% and increase in LV volumes according to echocardiography (ECHO)
  Exclusion criteria:
  1. Presence of contraindications to the stress test with inotropic stimulation;
  2. inflammatory myocardial diseases;
  3. the presence of severe hematological, neurological disorders, other psychosomatic conditions that impede research;
  4. life expectancy of less than 6 months (acute renal and hepatic failure, mental illness, malignant neoplasms of the final stages, unsuitable correction of brain injury).
  Interventions: Diagnostic Test: Stress Gated blood pool SPECT
- Ischemic cardiomyopathy group - 2 (ICM-2): Inclusion criteria:
  1. History of myocardial infarction (MI) or revascularization (CABG or PCI);
  2. > 75% stenosis of left main or proximal LAD and/ or stenosis of > 75% of ≥2 epicardial vessels (based on coronary angiography (CA) data);
  3. LV EF <40% and increase in LV volumes according to echocardiography (ECHO)
  Exclusion criteria:
  1. Presence of contraindications to the stress test with inotropic stimulation;
  2. inflammatory myocardial diseases;
  3. the presence of severe hematological, neurological disorders, other psychosomatic conditions that impede research;
  4. life expectancy of less than 6 months (acute renal and hepatic failure, mental illness, malignant neoplasms of the final stages, unsuitable correction of brain injury).
  Interventions: Diagnostic Test: Dynamic SPECT
- Control group for GBPS.: Inclusion criteria:
  1. Absence of obstructive coronary artery lesion;
  2. Absence of history of MI and revascularization.
  Exclusion criteria:
  1. Presence of contraindications to the stress test with inotropic stimulation;
  2. inflammatory myocardial diseases;
  3. the presence of severe hematological, neurological disorders, other psychosomatic conditions that impede research;
  4. life expectancy of less than 6 months (acute renal and hepatic failure, mental illness, malignant neoplasms of the final stages, unsuitable correction of brain injury).
  Interventions: Diagnostic Test: Stress Gated blood pool SPECT
- Control group for CFR.: 1. Presence of obstructive coronary artery lesion;
  2. Indications for coronary artery bypass grafting
  Exclusion criteria:
  1. Presence of contraindications to the adenosine stress test;
  2. inflammatory myocardial diseases;
  3. the presence of severe hematological, neurological disorders, other psychosomatic conditions that impede research;
  4. life expectancy of less than 6 months (acute renal and hepatic failure, mental illness, malignant neoplasms of the final stages, unsuitable correction of brain injury).
  Interventions: Diagnostic Test: Dynamic SPECT

INTERVENTIONS:
Diagnostic Test: Stress Gated blood pool SPECT — After labeling of red blood cells in vivo, a sequential series of acquisition is carried out at rest and during increasing doses of dobutamine (5/10/15 μg / kg / min). The duration of acquisition is 300 seconds.
  The acquisitions are carried out on dedicated cardiac gamma-camera with ultrafast Cadmium zinc telluride (CZT) detectors (DiscoveryNM530c, General electric Healthcare Israel, Israel)
  Other Names: Stress radionuclide angiography; Stress radionuclide ventriculography
  Groups: Control group for GBPS.; Ischemic cardiomyopathy group - 1 (ICM-1)
Diagnostic Test: Dynamic SPECT — The passage of a radiopharmaceutical bolus through the cavities of the heart and myocardium at rest and during infusion of adenosine at a dosage of 140 mcg / kg / min (for 4 minutes) is recorded.
  At the peak of the stress test (after 2 minutes of administration of adenosine), a 5 ml bolus (dose 260-444 MBq) of 99mTc-methoxyisobutylisonitrile (MIBI) is administered at a rate of 1 ml / s. Immediately after the end of tracer administration, 30 ml of 0.9% sodium chloride (NaCl) is infused. A scintigraphic recording of the study begins 5 seconds before the administration of the radiopharmaceutical.
  The next day, the study at rest is carried out. Scintigraphic images are recorded in tomographic mode with ECG synchronization for 600 s, at list mode.
  The acquisitions are carried out on dedicated cardiac gamma-camera with ultrafast CZT detectors (DiscoveryNM530c, General electric Healthcare Israel, Israel)
  Other Names: Radionuclide coronary flow reserve assessement
  Groups: Control group for CFR.; Ischemic cardiomyopathy group - 2 (ICM-2)

SUMMARY:
According to single-photon emission computed tomography, the left ventricular contractile and coronary flow reserve (CFR) will be assessed in patients with ischemic cardiomyopathy. According to these data, the criteria for predicting the effectiveness of complex surgical treatment of this pathology will be evaluated.

DETAILED DESCRIPTION:
Before surgical intervention, all patients pass routine clinical analyzes undergo coronary angiography and 2D echocardiography. Some of patients in the ICM-1 and ICM-2 groups undergo stress echocardiography with dobutamine.

Coronary arteriography is performed using the Axiom Artis (Siemens; Erlangen, Germany) and transthoracic two-dimensional Doppler echocardiography (TTE) with the Acuson Sequoia 512 (Siemens; Erlangen, Germany)).

Besides, all of the ICM-1 and ICM-2 groups patients undergo myocardial perfusion imaging. Standard two-day stress-rest imaging protocol is used. Adenosine at a dosage of 140 mcg/kg/min (for 4 min) is used as a pharmaceutical stress agent.

ICM-1 group and Control group for GBPS undergo gated blood pool SPECT (GBPS) at rest and during increasing doses of dobutamine (5/10/15 μg/kg/min) (n = 60) ICM-2 group and Control group for CFR undergo dynamic SPECT (n = 40). This investigation is combined with routine myocardial perfusion imaging so patients are not exposed to extra stress.

Than ICM patients undergo surgical treatment of ICM in different volume. All of them receive coronary bypass grafting (CABG); some patients undergo the left ventricular reconstruction and intervention on the mitral valve.

In the early postoperative period (7-14 days), the ICM-1 group undergo rest GBPS and ICM-2 group undergo dynamic SPECT by two-day protocol. All patients undergo TTE too.

After at least 12 month, all patients undergo TTE to assess the presence of left ventricular (LV) remodeling.

ELIGIBILITY:
Inclusion Criteria:

А) For ICM group:

1. History of myocardial infarction (MI) or revascularization (CABG or PCI);
2. > 75% stenosis of left main or proximal LAD and/ or stenosis of > 75% of ≥2 epicardial vessels (based on coronary angiography (CA) data);
3. LV EF <40% and increase in LV volumes according to echocardiography (ECHO)

B) For GBPS Control group

1. Absence of obstructive coronary artery lesion;
2. Absence of history of MI and revascularization.

C) For CFR Control group

1. Presence of obstructive coronary artery lesion;
2. Indications for coronary artery bypass grafting;

Exclusion Criteria (for all groups):

1. Presence of contraindications to the stress test with inotropic stimulation;
2. Inflammatory myocardial diseases;
3. The presence of severe hematological, neurological disorders, other psychosomatic conditions that impede research;
4. Life expectancy of less than 6 months (acute renal and hepatic failure, mental illness, malignant neoplasms of the final stages, unsuitable correction of brain injury).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being living in Russian Federation (inc.ethnic minorities)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an ongoing LV remodeling and reverse LV remodeling. | 12 month
  Ongoing LV remodeling is meant increase of LV end-systolic volume (LVESV) or decrease of LVESV≤10% according to 2D echocardiography in comparison to early postoperative period study. Reverse LV remodeling is meant decrease in LVESV >10% according to 2D echocardiography in comparison to early postoperative period study.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Zavadovsky, MD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Centre
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Centre, Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shipulin VV, Andreev SL, Pryakhin AS, Mochula AV, Maltseva AN, Sazonova SI, Shipulin VM, Massalha S, Zavadovsky KV. Low-dose dobutamine stress gated blood pool SPECT assessment of left ventricular contractile reserve in ischemic cardiomyopathy: a feasibility study. Eur J Nucl Med Mol Imaging. 2022 Jun;49(7):2219-2231. doi: 10.1007/s00259-022-05714-y. Epub 2022 Feb 12. PMID 35150293